CLINICAL TRIAL: NCT00442338
Title: MK-476 IV Formulation Phase III Open Label Exploratory Comparative Study - Acute Exacerbations of Asthma -
Brief Title: Study of MK-0476 in Adult Patients With Acute Asthma (0476-334)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0476-334; MK-0476-334; 2007_007
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Results first posted 2009-07-14 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast; Theophylline

ARMS (3):
- Montelukast 7 mg (Experimental): Montelukast 7 mg IV administration
  Interventions: Drug: montelukast sodium
- Montelukast 14 mg (Experimental): Montelukast 14 mg IV administration
  Interventions: Drug: montelukast sodium
- Aminophylline 250 mg (Active Comparator): Aminophylline 250 mg IV drip administration
  Interventions: Drug: aminophylline hydrate

INTERVENTIONS:
Drug: montelukast sodium — Montelukast 7 mg single injection (IV bolus administration) over 2-3 minutes
  Other Names: MK-0476
  Arms: Montelukast 7 mg
Drug: montelukast sodium — Montelukast 14 mg single injection (IV bolus administration) over 5 minutes
  Other Names: MK-0476
  Arms: Montelukast 14 mg
Drug: aminophylline hydrate — Aminophylline 250 mg IV drip infusion over 60 minutes
  Other Names: Kyophyllin® Injection 2.5%, FK05
  Arms: Aminophylline 250 mg

SUMMARY:
The study estimates the efficacy and safety of MK0476 and aminophylline intravenous administration in adult participants with acute asthma.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants with acute asthma attacks

Exclusion Criteria:

* Participant has any known or suspected, acute or chronic cause for their pulmonary symptoms other than asthma (e.g., COPD, chronic heart failure, etc.).
* Participant has a smoking habit (15 cigarettes per day) within a month prior to screening period, and/or has a smoking history (20 cigarettes per day) of more than 15 years.
* Participant has a disease of the cardiovascular, hepatic, renal, hematologic systems, or other severe disease.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2007-03; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III.
  Studied period: March 12, 2007 (date study drug was first administered to first participant) to August 1, 2007 (date study drug was last administered to last participant). Study was conducted at 31 clinical sites.
Pre-assignment Details: Participants with acute exacerbation of bronchial asthma received standard treatments of inhaled β-agonist or oxygen inhalation to treat the acute exacerbations during the 60 minutes in the screening period before the study randomization.
Groups:
- Montelukast 14 mg: Montelukast 14 mg Intravenous Administration
Period: Overall Study
Arm/Group | Montelukast 7 mg | Montelukast 14 mg | Aminophylline 250 mg
Started | 30 | 30 | 31
Completed | 30 | 30 | 31
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast 7 mg | Montelukast 14 mg | Aminophylline 250 mg | Total
Number analyzed (Participants) | 30 | 30 | 31 | 91
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.0 (12.3) | 56.7 (15.2) | 55.4 (14.5) | 56.0 (13.9)
Age, Customized [Number; unit: Participants]
  Adolescents (12-17 years) | 0 (12.3) | 1 (15.2) | 0 (14.5) | 1
  Adults (18-64 years) | 21 | 16 | 20 | 57
  From 65-84 years | 9 | 13 | 11 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 16 | 62
  Male | 8 | 6 | 15 | 29
Asthma Attack Severity based on Asthma Prevention and Management Guideline 2003, Japan [Number; unit: Participants] — Mild (Peak Expiratory Flow: 70%-80%), Moderate (Peak Expiratory Flow: 50%-70%), Severe (Peak Expiratory Flow: <=50%) or Serious (Peak Expiratory Flow: incapable measurement, cyanosis, head trip, disturbed consciousness, incontinence or asphyxia)
  Participants
    Mild | 21 (0.29) | 18 (0.33) | 26 (0.53) | 65
    Moderate | 9 | 12 | 5 | 26
    Severe | 0 | 0 | 0 | 0
    Serious | 0 | 0 | 0 | 0
Baseline Forced Expiratory Volume in One Second (FEV1) [Mean (Standard Deviation); unit: Liter] | 1.35 (0.29) | 1.18 (0.33) | 1.43 (0.53) | 1.32 (0.41)
Duration of Asthma [Mean (Standard Deviation); unit: Years] | 14.9 (10.4) | 13.9 (11.5) | 16.7 (14.1) | 15.2 (12.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1) Within the First 60 Minutes After Administration
Description: The time weighted average change from Baseline in Forced Expiratory Volume in One Second (FEV1) over the first 60 minutes after study drug administration (average change FEV1 (0-60 min)). Baseline (pre-allocation) was the last measurement obtained during the screening period.
Time Frame: Baseline and 60 minutes after study drug administration
Population: Per Protocol Set (PPS): subset of participants who comply with the protocol sufficiently to ensure that these data will likely exhibit effects of treatment, according to the underlying scientific model. Aminophylline 250 mg - 1 participant with no FEV1 data at 60 minutes was excluded from the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | Montelukast 7 mg | Montelukast 14 mg | Aminophylline 250 mg
Number analyzed (Participants) | 27 | 30 | 29
Liter | 0.07 [0.02 to 0.12] | 0.05 [0.00 to 0.11] | 0.06 [0.01 to 0.12]
Statistical Analysis 1: Comparison: Montelukast 7 mg vs Aminophylline 250 mg; Treatment difference in change from Baseline in FEV1 within the first 60 minutes after study drug administration was assessed as the difference in the least square (LS) means of time weighted average change FEV1 (0-60 min) using an Analysis of Covariance (ANCOVA) model; Test type: Superiority or Other; p = 0.871, ANCOVA; The model included a factor for treatment and used the baseline FEV1 as a covariate; Difference in LS Means = 0.01, 95% CI 2-sided [-0.07 to 0.08]
Statistical Analysis 2: Comparison: Montelukast 14 mg vs Aminophylline 250 mg; Treatment difference in change from Baseline in FEV1 within the first 60 minutes after study drug administration was assessed as the difference in the LS means of time weighted average change FEV1 (0-60 min) using an ANCOVA model; Test type: Superiority or Other; p = 0.794, ANCOVA; The model included a factor for treatment and used the baseline FEV1 as a covariate; Difference in LS Means = -0.01, 95% CI 2-sided [-0.08 to 0.06]
Statistical Analysis 3: Comparison: Montelukast 7 mg vs Montelukast 14 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.675, ANCOVA; The model included a factor for treatment and used the baseline FEV1 as a covariate; Difference in LS Means = 0.02, 95% CI 2-sided [-0.06 to 0.09]

ADVERSE EVENTS:
Time Frame: From Screening through post-trial visit (up to 14 days)
Arm/Group | Montelukast 7 mg | Montelukast 14 mg | Aminophylline 250 mg
Serious Adverse Events (participants affected / at risk) | 3/30 | 0/30 | 1/31
Other Adverse Events (participants affected / at risk) | 5/30 | 1/30 | 3/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Montelukast 7 mg (N=30) | Montelukast 14 mg (N=30) | Aminophylline 250 mg (N=31)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Montelukast 7 mg (N=30) | Montelukast 14 mg (N=30) | Aminophylline 250 mg (N=31)
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 0
Glucose urine present (Investigations) | 2 | 1 | 1
Oedema (General disorders) | 2 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.